CLINICAL TRIAL: NCT06910891
Title: Hemodynamic Evaluation Using Microcirculation for Early Treatment of Septic Patients
Acronym: HEMOCAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87RI24_0047 (HEMOCAP; 2025-A00216-43 (Other: IDRCB)
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Emergency Care; Microcirculation
Keywords: microcirculation; septic patient; organ dysfunction; sepsis; peripheral perfusion index; emergency unit
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Intervention Model Description: Quasi-experimental interventional study of the here-elsewhere type, open and multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): As soon as an eligible patient is identified by the nurse, in addition to the classic hemodynamic parameters measured in all patients, a measurement of the peripheral perfusion index (from 1 sec to 10 sec) and marbling assessment (scale from 0 to 5) will be performed. This measurement will be validated by the senior doctor of the Sepsis Department. When the peripheral perfusion index will be ≥ 3 sec and/or the marbling score ≥ 1, a first vascular filling test of 500 cc over 30 minutes will be started, regardless of the value of the hemodynamic parameters.
  Interventions: Diagnostic Test: measurement of the peripheral perfusion index and marbling assessment
- Control arm (No Intervention): Patients will benefit from treatment according to current standards of care

INTERVENTIONS:
Diagnostic Test: measurement of the peripheral perfusion index and marbling assessment — in addition to the classic hemodynamic parameters measured in all patients, a measurement of the peripheral perfusion index (from 1 sec to 10 sec) and marbling assessment (scale from 0 to 5) will be performed
  Arms: Intervention arm

SUMMARY:
Despite early treatment, the deterioration and mortality of sepsis patients remains high. A possible explanation could be persistent tissue hypoperfusion, or undetected in the early phase despite the normalization of macro-hemodynamic parameters. This interventional study evaluates the impact of measuring microcirculation parameters by nurses on patient prognosis through early initiation of vascular filling.

DETAILED DESCRIPTION:
Sepsis and its most serious form, septic shock, are a public health problem. Sepsis is defined by the presence of organ failure, including acute circulatory failure, which combines hypovolemia, vasoplegia and cardiac dysfunction. Vascular filling is therefore a pillar of the management of septic patients to correct hypovolemia and improve perfusion and tissue oxygenation. Following numerous studies, the evaluation of peripheral microcirculation is becoming a clinical "trigger" making it possible to identify patients at risk, particularly in emergency department. In a meta-analysis, it has been showed that alterations in microcirculatory perfusion predict deterioration and mortality during severe infections. Currently, no interventional study has evaluated the impact of measuring microcirculatory perfusion (peripheral perfusion index and marbling) by nurses on patient prognosis through early initiation of vascular filling.

In this study, patients will be assessed hemodynamically using peripheral perfusion index and/or presence of mottling. If peripheral perfusion index > 3s and/or presence of marbling a first vascular filling test of 500 cc over 30 minutes will be started after a medical control.

Patient will be followed up 7 days to determine outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Admitted to the Emergency Department for suspected Sepsis for less than 6 hours according to international Sepsis-3 definitions (high probability of infection defined by a fever greater than or equal tol to 38.3°C with a suspected infectious source + Score NEWS 2 greater than or equal to 2)
3. Affiliated to a social security system
4. Having agreed to participate in this study

Exclusion Criteria:

1. Patient with arterial hypotension (SBP ≤ 100 mmHg) on admission
2. Patient having already received a 500mL filling test over 30 minutes
3. Patients moribund according to the investigator
4. Pregnancy or breastfeeding
5. Patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of patients presenting clinical deterioration during emergency care | between time of inclusion and 24 hours after
  Clinical deterioration is defined by (composite criterion):
  1. Arterial hypotension defined by systolic blood pressure (SBP) ≤ 100 mmHg
  2. Implementation of treatment for organ support:
     * Vasopressor or inotrope
     * Invasive ventilation
  3. Abnormal lactate concentration (> 2mmol/L), without improvement (absence of decay)
  4. Patient admitted in intensive care unit
  5. Death

SECONDARY OUTCOMES:
Number and proportion of patients who received bundles (i) one hour and (ii) 3 hours of admission to the Emergency Department | from admission to the Emergency Department to 3 hours after
Difference in SOFA score (≥ 2 points) between Hours 0 and Hours 24 (24h±6h) | between Hours 0 and Hours 24
Number and proportion of deaths on Day 7 | from enrollement to the end of the patient participation at Day 7
Number and proportion of patients with hydrostatic pulmonary oedema (cardiogenic or volume overload) or receiving diuretic treatment during emergency care | from enrollment to the end of the subject participation at day 7
The correlation of the peripheral perfusion index measurement (pathological : yes/no) between the nurse and the emergency physician | hour 0
Number and proportion of patients sent home, conventional hospitalization or intensive care | from enrollment to the end of the subject participation at day 7

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Brive Hospital, Brivé
  - Guéret Hospital, Guéret
  - Limoges University Hospital, Limoges
  - Saint Junien Hospital, Saint-Junien
  - Tulle Hospital, Tulle
  - Ussel Hospital, Ussel